CLINICAL TRIAL: NCT01392105
Title: A Randomized, Open-label, Multicenter Trial for the Safety and Efficacy of Intracoronary Adult Human Mesenchymal Stem Cells After Acute Myocardial Infarction
Brief Title: Safety and Efficacy of Intracoronary Adult Human Mesenchymal Stem Cells After Acute Myocardial Infarction
Acronym: SEED-MSC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: FCB-Pharmicell Co Ltd. (Unknown)
Responsible Party: Seung-Hwan Lee/Professor, Yonsei University Wonju College of Medicine, Wonju Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC2-Version 6.0
Record Dates: First submitted 2011-07-05; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Mesenchymal stem cells; Myocardial infarction; Left ventricular dysfunction
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell treatment group (Active Comparator)
  Interventions: Drug: Mesenchymal stem cell
- Control group (Placebo Comparator): All patients were required to have successful revascularization of an infarct-related artery on coronary angiography at the time of randomization. All patients received aspirin (300 mg loading dose, then 100 mg daily) and clopidogrel (600 mg loading dose, then 75 mg daily) with optimal medical therapy according to the American College of Cardiology (ACC)/ American Heart Association (AHA) guidelines for treatment of ST-segment elevation myocardial infarction (STEMI)
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Mesenchymal stem cell — Route : intracoronary injection Frequency : single dose of autologous bone-marrow derived mesenchymal stem cells Dosage : 1x1000000 cells/kg Duration : mean injection duration approximately 4 weeks after primary percutaneous coronary intervention
  Other Names: Hearticellgram-AMI
  Arms: Mesenchymal stem cell treatment group
Drug: Control group — No additional treatment of mesenchymal stem cells
  Arms: Control group

SUMMARY:
Early reperfusion strategies in tandem with remarkable advances in drugs and devices for treating myocardial infarction (MI) have contributed to a reduction in early mortality, but cardiovascular disease remains the leading cause of death worldwide. Current management strategies cannot solve the problem of cardiomyocyte loss and consequent progression of heart failure. In this respect, stem-cell therapy has shown potential benefits for repairing the damaged myocardium. Mesenchymal stem cells (MSCs) have been considered to be attractive therapeutic candidates because of their high capacity for replication: paracrine effect: ability to preserve potency: and because they do not cause adverse reactions to allogeneic versus autologous transplants. Intracoronary injection of stem cells seems to be safe, but only one clinical trial using MSCs via the intracoronary route in the setting of acute myocardial infarction (AMI) has been carried out. The investigators therefore assessed the safety and efficacy of intracoronary autologous bone marrow (BM)-derived human MSCs in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years
* ischemic chest pain for >30 min
* admitted to hospital <24 h after the onset of chest pain
* electrocardiography showed ST segment elevation >1 mm in two consecutive leads in the limb leads or >2 mm in the precordial leads
* they could be enrolled in the study <72 h after successful revascularization

Exclusion Criteria:

* cardiogenic shock (defined as systolic blood pressure <90 mmHg requiring intravenous pressors or intra-aortic balloon counterpulsation)
* life-threatening arrhythmia
* impossible conditions for cardiac catheterization
* advanced renal or hepatic dysfunction
* history of previous coronary artery bypass graft
* history of hematologic disease
* history of malignancy
* major bleeding requiring blood transfusion
* stroke or transient ischemic attack in the previous 6 months
* structural abnormalities of the central nervous system (brain tumor, aneurysm, history of surgery)
* traumatic injury after myocardial infarction
* use of corticosteroids or antibiotics during the previous month
* major surgical procedure in the previous 3 months
* cardiopulmonary resuscitation for >10 min within the previous 2 weeks
* positive skin test for penicillin
* positive result for viral markers (human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and Venereal Disease Research Laboratory (VDRL) test)
* pregnancy, possible candidate for pregnancy or breastfeeding females
* drug abusers
* inappropriate patients to participate in the study according to the chief investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Absolute changes in global LVEF by SPECT | baseline and 6 months
  Absolute changes in global left ventricular ejection fraction (LVEF) as measured by SPECT 6 months after cell infusion

SECONDARY OUTCOMES:
Changes in left ventricular end-diastolic volume (LVEDV) | baseline and 6 months
Changes in left ventricular end-systolic volume (LVESV) | baseline and 6 months
Changes in regional wall motion score index (WMSI) by Echocardiography | baseline and 6 months
Major adverse cardiac event (MACE) | 6 months
  MACE was defined as the composites of any cause of death, myocardial infarction, revascularization of the target vessel, re-hospitalization for heart failure, and life-threatening arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Yonsei University Wonju College of Medicine, Wonju Christian Hospital
Locations (3):
- South Korea (3):
  - Yonsei University Wonju College of Medicine, Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Inha University Hospital, Inchon
  - Yonsei Cardiovascular Center and Cardiovascular Research Institute, Yonsei University College of Medicine, Seoul

REFERENCES:
- [Derived] Lee JW, Lee SH, Youn YJ, Ahn MS, Kim JY, Yoo BS, Yoon J, Kwon W, Hong IS, Lee K, Kwan J, Park KS, Choi D, Jang YS, Hong MK. A randomized, open-label, multicenter trial for the safety and efficacy of adult mesenchymal stem cells after acute myocardial infarction. J Korean Med Sci. 2014 Jan;29(1):23-31. doi: 10.3346/jkms.2014.29.1.23. Epub 2013 Dec 26. PMID 24431901